CLINICAL TRIAL: NCT01003223
Title: Phosphate Kinetic Modeling
Acronym: PKM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEIRB PKM 09-207
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2010-11

CONDITIONS: End Stage Renal Disease; Hyperphosphatemia
Keywords: phosphorus; dialysis; PhosLo; CKD stage V
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PKM modeling with graphical report (Experimental)
  Interventions: Other: Computer algorithm management of hyperphosphatemia

INTERVENTIONS:
Other: Computer algorithm management of hyperphosphatemia — The PKM algorithm is a computer based program that calculates Phosphorus intake between dialysis, phosphorus reduction during dialysis treatment and daily oral phosphate binder intake compliance. Based on pre and post dialysis serum phosphorus levels, the algorithm makes recommendations in relation to dialysate calcium, oral phosphate binder use, and dietary counseling.

SUMMARY:
Cardiovascular disease is a major cause of death in hemodialysis (HD) patients and is associated with widespread vascular calcification. There is a consensus that the chronic overload of calcium and phosphorus is a major factor in vascular calcification. Hyperphosphatemia, deleterious in dialysis patients, is aggressively monitored and treated. Phosphate binders - designed to bind dietary phosphate and thus prevent its absorption, are ubiquitous in the dialysis patient population, and calcium-based phosphate binders are often first line therapy because they are tolerated well by the patients and low in cost. Phosphate Kinetic Modeling (PKM) is a tool to help physicians manage a hemodialysis patient's phosphate level. Once a subject consents to participate in the study, the subject's dietary phosphate intake will be estimated and the appropriate dose of the phosphate binder calcium acetate (PhosLo) will be recommended accordingly. If necessary, the Ca++ concentration of the dialysate will be changed to remove any excess calcium absorbed as the result of an increase in the PhosLo prescription to control phosphorus.Ongoing recommendations regarding oral phosphate binders dialysate calcium will be made using a computer generated algorithm.

DETAILED DESCRIPTION:
PKM consists of a set of validated and computerized algorithms to perform the following steps:

1. Calculate calcium (Ca) and phosphorus (P) intake and absorption in individual patients as a function of the prescribed doses of Vitamin D analogues, protein catabolic rate (PCR) and dietary and binder Ca intakes.
2. Calculate P removal between dialyses by P binders and P and Ca removal during dialysis from kinetic analysis of total P and Ca transport during dialysis based on dialyzer P and Ca transport coefficients and the levels of dialysate Ca and serum Ca and P.
3. Thus from analysis of intake, absorption and removal the program can calculate net Ca and P balance in modeled patients.
4. Calculate the dose of phosphate binder required to reduce the serum P to normal in patients with hyperphosphatemia.
5. Calculate the dialysate Ca required to achieve zero calcium balance over complete dialysis cycles - the interdialytic interval and immediately succeeding dialytic interval.
6. The program also computes a Phosphorus-Protein index (PPI, the total P removed divided by PCR, mg/gm/day) which provides a quantitative index of compliance with prescribed dietary P restriction and/or the prescribed dose of binders. If the PPI exceeds 18, the report indicates it is likely the patient is not in compliance with respect to prescribed diet and/or binder. It is hoped that this information will be valuable to guide semiquantitative evaluations of diet P and binder intakes in patients difficult to manage.

Patients will be modeled on a monthly basis from pre- and post-dialytic Ca, P, PCR and other routine data readily available such as blood and dialysate flow rates, fluid removal etc. A monthly report will be generated for the physician and staff by Norma Ofsthun, PhD containing the analyses and recommendations for any changes in therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Thrice weekly hemodialysis with a dialysate Ca++ concentration (CdiCa) of 2.25 or 2.5 mEq/L
3. Stable CdiCa of either 2.25 or 2.5 mEq/L for ≥ 4 weeks
4. Dialysis vintage ≥ 6 months
5. Current serum phosphorus ("month -1") > 5.5 mg/dL and average serum phosphorus month -1 to -3 > 5.5 mg/dL and average serum phosphorus month -1 to -6 > 5.5 mg/dL
6. Patients currently prescribed calcium acetate (PhosLo) mono-therapy , sevelamer monotherapy, or a combination therapy of PhosLo plus sevelamer for phosphate binding
7. Fresenius Optiflux F 160, 180 or 200 dialyzer

Exclusion Criteria:

1. Parathyroidectomy
2. iPTH < 50 pg/mL
3. Dialysate potassium prescription other than 2 or 3 mmol/L Corrected serum Ca++ < 7.5 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is the change in serum phosphorus between a baseline period and the final 4 months of the study period. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fresenius Medical Services, Waltham, Massachusetts, United States